CLINICAL TRIAL: NCT01625637
Title: Tobacco Approach Avoidance Training for A Smoking Cessation in Adolescent Smokers- Study 2
Brief Title: Tobacco Approach Avoidance Training for Adolescent Smokers-2
Acronym: AAT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1103008127-2
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-08

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine; Smoking; Adolescent; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AAT-avoid cigarette condition (Experimental): Adolescent smokers are trained to avoid tobacco in a training AAT
  Interventions: Behavioral: AAT-experiment
- AAT-no contingency continued assessment (Placebo Comparator)
  Interventions: Behavioral: AAT-placebo

INTERVENTIONS:
Behavioral: AAT-experiment — This AAT condition trains kids to avoid cigarettes
  Arms: AAT-avoid cigarette condition
Behavioral: AAT-placebo — This AAT condition is a no contingency continued assessment version (50% approach-cigarettes, 50% avoid cigarettes).
  Arms: AAT-no contingency continued assessment

SUMMARY:
This is a two part study. In Study 2, smokers who want to quit smoking will participate in a 4 week smoking cessation program combining weekly cognitive behavioral therapy (CBT) with weekly regular-AAT or placebo-AAT training. We hypothesize that adolescent smokers will exhibit stronger approach tendencies towards smoking-related stimuli in the tobacco Approach Avoidance Training (AAT) task when compared with nonsmokers and that adolescent smokers who are trained to avoid smoking related stimuli using the AAT will avoid tobacco approach tendencies in the AAT test trials and the Implicit Association Task, when compared to adolescent smokers who are not exposed to AAT training. We also hypothesize that adolescent smokers who are trained to avoid tobacco in a training AAT in combination with CBT will have better abstinence rates compared to those who receive placebo AAT training with CBT.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Between ages 13-18 years
* Able to read and write in English.
* Smokers: Smoking 5 or more cigarettes daily for at least 6 months; Baseline urine cotinine levels > 500 ng/ml
* Nonsmokers: Never smokers; Baseline urine cotinine levels < 50 ng/ml

Exclusion Criteria:

* Current criteria for dependence on another psychoactive substance
* Current diagnosis of psychosis, major depression or panic disorder
* Regular use of any psychoactive drugs including anxiolytics and antidepressants unless the medication has been taken consistently for 2 months, is currently being monitored by a physician, and the condition for which the medication is taken is considered to be stable
* Pregnant or lactating girls, based on self report.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked | 4 weeks
  To evaluate if retraining automatic approach tendencies towards smoking stimuli, in combination with CBT, enhances an adolescent's ability to quit smoking following 4 weeks of treatment for smoking cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, School of Medicine, Department of Psychiatry, New Haven, Connecticut, United States